CLINICAL TRIAL: NCT00362245
Title: Amikacin Penetration Into the Cerebrospinal Fluid: Pharmacokinetic/Pharmacodynamic Analysis in Adults With Hospital Acquired Gram-negative Meningitis Associated With Intracranial Pressure Monitoring and Draining Devices
Brief Title: Amikacin Penetration Into the Cerebrospinal Fluid
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of participants
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07/2006_CTIL
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Gram Negative Meningitis; Post Traumatic Bacterial Meningitis
Keywords: Amikacin; Pharmacokinetics; Pharmacodynamics; Intra-Thecal injection

INTERVENTIONS:
Drug: Systemic and Intra-Thecal Amikacin Therapy

SUMMARY:
The limited available data precludes establishing an antibiotic regimen in patients suffering from bacterial meningitis after head trauma, or spontaneous bleeding Understanding the disposition of Amikacin administered intrathecally will enable to propose rational treatment of these patients.

DETAILED DESCRIPTION:
The limited available data precludes establishing an antibiotic regimen in patients suffering from bacterial meningitis after head trauma, or spontaneous bleeding Understanding the disposition of Amikacin administered intrathecally will enable to propose rational treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Culture proved bacterial meningitis where the prescribed therapy includes the use of systemic and intraventricular amikacin therapy.
2. The included patient should have an intraventricular catheter placed for intraventricular pressure measurement and admitted to an intensive care unit.
3. Blood creatinine concentration up to 1.49 mg/dL measured at the inclusion day.

Exclusion Criteria:

1. Patients or legal guardians who refuse to participate in the study.
2. Known allergy to amikacin.
3. Blood creatinine concentration of 1.5 mg/dL or higher.
4. Subjects without intraventricular catheter who will need repeated lumbar punctures for CSF amikacin determinations.
5. Patients suffering from known chronic liver disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Bactericidal effect on the causative bacteria
Blood and CSF AUC/MIC relationship

CONTACTS AND LOCATIONS:
Overall Officials: Yedidiah Bentur, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel